CLINICAL TRIAL: NCT00699296
Title: A Phase II Study of Oral LBH589 in Patients With Cutaneous T-cell Lymphoma and Adult T-cell Leukemia/Lymphoma
Brief Title: Study of Oral LBH589 in Patients With Cutaneous T-cell Lymphoma and Adult T-cell Leukemia/Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B1201
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Cutaneous T-Cell Lymphoma; Leukemia-Lymphoma, Adult T-Cell
Keywords: LBH589; HDAC inhibitor; cutaneous T-ceII lymphoma; adult T-cell leukemia
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Leukemia-Lymphoma, Adult T-Cell | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Panobinostat (LBH589)

INTERVENTIONS:
Drug: Panobinostat (LBH589) — 20mg/day p.o. on three times-a- week
  Other Names: LBH589

SUMMARY:
This study will assess the safety, efficacy and pharmacokinetics of oral LBH589 in Japanese adult patients with refractory cutaneous T-Cell Lymphoma and adult T-cell leukemia/lymphoma. LBH589 is administered orally once a day for three days per week.

ELIGIBILITY:
Inclusion criteria:

* CTCL: Biopsy-confirmed MF or SS stages IB-IVA2.
* Patients who have SS with bone marrow involvement are also eligible.
* Patients with transformed CTCL are eligible.
* ATL: Patient with cytologically or histopathologically confirmed lymphoma.
* Lymphoma should be identified as tumors derived peripheral T-cells by cell surface marker.
* ATL: Patients with positivity for anti-HTLV-1 antibody
* Patients must have received at least two systemic therapy regimens.
* Patients must have had disease progression on or following their most recent treatment regimen.
* Age ≥ 20 years
* ECOG Performance Status of ≤ 2
* Written informed consent obtained prior to any study specific screening procedures

Exclusion criteria:

* Patients with a history of primary CNS tumors
* Any history or presence of brain metastases
* Patients with any peripheral neuropathy ≥ CTCAE grade 2
* Patients with unresolved diarrhea > CTCAE grade 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
* Patients with concurrent severe and/or uncontrolled liver or renal disease
* Patients using sodium valproate ≤5 days prior to starting study drug
* Patients with an active bleeding diathesis or on any treatment with therapeutic doses of sodium warfarin or other antivitamin K drugs
* Patients who have received any investigational drug or chemotherapy or undergone major surgery ≤ 3 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have received biologic therapy, target therapy (e.g. denileukin diftitix ), vaccine, systemic steroids or immunotherapy ≤ 2 weeks prior to starting study treatment or who have not recovered from side effects of such therapy
* Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Overall response (CR/PR) rate by using the modified Severity-Weighted Assessment Tool (mSWAT) to assess skin disease and the combined evaluation of disease in the viscera/lymph nodes, peripheral blood and bone marrow | Every Cycle

SECONDARY OUTCOMES:
Response rate using mSWAT Response rate using the Physician's Global Assessment of Clinical Condition (PGA) Responses in index lesions by skin lesion measurements and with photographic supporting documentation Overall response(CR/PR) rate by using PG | 1 cycle

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Sugaya, Principal Investigator — The University of Tokyo Hospital; Kenji Iwatsuki, Principal Investigator — Okayama University; Yoshiki Tokura, Principal Investigator — University Hospital of Occupational and Environmental Health; Kunihiro Tsukasaki, Principal Investigator — Nagasaki University Hospital of Medicine and Dentistry; Hironobu In, Principal Investigator — Kumamoto University Hospital; Mitsuru Setoyama, Principal Investigator — University of Miyazaki Hospital; Atae Utsunomiya, Principal Investigator — Imamura Bun-in Hospital
Locations (7):
- Japan (7):
  - University Hospital of Occupational and Environmental Health, Fukuoka
  - Imamura Bun-in Hospital, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - University of Miyazaki Hospital, Miyazaki
  - Nagasaki University Hospital of Medicine and Dentistry, Nagasaki
  - Okayama University Hospital, Okayama
  - The University of Tokyo Hospital, Tokyo